CLINICAL TRIAL: NCT04815369
Title: Evaluating UTI Diagnosis in Nursing Homes
Status: Withdrawn | Type: Observational
Why Stopped: No Enrollment
Sponsor: Pathnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-PUTINH
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2024-11

CONDITIONS: Urinary Tract Infections
Keywords: Nursing Home; Clostridium difficile; PCR; Long Term Care Facility; Skilled Nursing Facility; National Healthcare Safety Network
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Guidance Clinical Pathway: Facilities will be provided a standardized infrastructure and process for collecting and reporting of urine test results including unique lab requisitions that contain the option to order Guidance® UTI, Standard Urine Culture (SUC), and Urine Analysis (UA) along with a protocol for results notification to a central point person within the Nursing Home (NH) facility
- Traditional Clinical Pathway: Facilities will employ their current standard clinical care practices for suspected UTI, including SUC, UA, and Guidance® UTI testing as per current reporting practices. Providers at these facilities will have the option to order any diagnostic test they deem appropriate.

SUMMARY:
This prospective, multicenter, comparative cohort observational study is to determine whether the use of Guidance® UTI Clinical Pathway, a standardized infrastructure for specimen collection and result delivery, compared with current traditional pathways for urine testing reduces the proportion of UTI patients with poor outcomes.

DETAILED DESCRIPTION:
The objective of this study is to determine if prospective data, collected over 12 months from over 200 nursing homes, will show that the use of Guidance® UTI Clinical Pathway is more effective than the Traditional Clinical Pathways for urine testing in UTI diagnosis in Nursing Homes. Guidance® UTI Clinical Pathway provides standardized infrastructure for specimen collection, and result dissemination via assigned report point person to verify receipt of actionable data. The pathway also includes several in-services on molecular testing for UTI, Pooled Antibiotic Susceptibility Testing, and polymicrobial infections to help providers better understand test methodology. Standardizing a Clinical Care Pathway for testing and reporting of clinical results approach may lead to a reduction in empiric broad spectrum antibiotic use and in turn better health-related outcomes for patients. Such efficiency in clinical decision making at the time of initial presentation may lead to improved patient care by avoiding ineffective therapy due to mismanagement or incomplete lab diagnosis. The study will be observing the implementation of the Guidance® UTI Clinical Pathway and comparing it to traditional clinical care pathways from facility-level data entered into the National Healthcare Safety Network for its LTCF (Long Term Care Facilities) Component.

ELIGIBILITY:
Inclusion

* Certified skilled nursing facilities (SNF) and nursing homes (NH)
* Nonprofit or for-profit freestanding facility certified by Medicare and Medicaid
* Currently utilizing an EMR system
* Minimum bed size of 100

Exclusion

* Assisted Living Facilities and Residential Care Facilities
* Participation in another UTI trial during the study period

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Cohort of residents residing in the NH facility during 12 consecutive months.-
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Examine prospective data to determine if the use of Guidance® UTI Clinical Pathway, compared to traditional clinical pathways, will reduce the proportion of patients with UTI-related adverse events. | 12 Months
  Examine the proportion of patients with UTI-related adverse events requiring emergency hospital services over the course the study with a composite measure of the number of UTI related ED visits and/or subsequent hospitalizations and/or sepsis events.

SECONDARY OUTCOMES:
Examine prospective data to determine if the use of Guidance® UTI Clinical Pathway, compared to traditional clinical pathways, will reduce overall inappropriate antibiotic use. | 30 Days
  Examine prospective data to determine if the use of Guidance® UTI Clinical Pathway, compared to traditional clinical pathways, will reduce overall inappropriate antibiotic use as measured by the rate of empiric antibiotic starts and the rate of antimicrobial changes for UTI indication.
Examine prospective data to determine if the use of Guidance® UTI Clinical Pathway is more effective than standard urine testing approaches in the clinical evaluation of UTI diagnosis and management . | 12 Months
  Examine prospective data to determine if the use of Guidance® UTI Clinical Pathway is more effective than standard urine testing approaches in the clinical evaluation of UTI diagnosis and management as measured by UTI incidence and corresponding urine testing rate
  * (UTI and Catheter associated (CA)-UTI bacterial identification incidence rates (diagnostic aim)
  * Population UTI Rate = (UTI Episodes/Resident Days) x 1,000
  * CA-UTI Rate = (CA-UTI Episode/Catheter days) x 1,000
Examine prospective data to determine if the use of Guidance® UTI Clinical Pathway, compared to traditional clinical pathways, will reduce UTI antibiotic collateral effects. | 30 Days
  Examine prospective data to determine if the use of Guidance® UTI Clinical Pathway, compared to traditional clinical pathways, will reduce UTI antibiotic collateral effects as measured by:
  * C. diff event rate = (Total C. diff events/ total resident days) x 1,000

CONTACTS AND LOCATIONS:
Overall Officials: Dave Baunoch, PhD, Principal Investigator — Clinical Trials
Locations (1):
- Pathnostics, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No